CLINICAL TRIAL: NCT03460431
Title: Evaluation of Fractional CO2 and Non Ablative Long Pulsed Nd YAG Lasers Alone and in Combination in Treatment of Keloids
Brief Title: A Study Using Fractional Carbon Dioxide and Long Pulsed Neodymium-yttrium Aluminum Garnet Lasers in Treatment of Keloids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Foad Mohamed, specialist of dermatology.students hospital. Cairo university, Cairo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3060114
Record Dates: First submitted 2018-01-23; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fractional CO2 laser 10,600nm (Experimental): fractional CO2 laser 10,600nm one session every month for 4 months
  Interventions: Device: fractional CO2 laser 10,600nm
- Nd YAG laser 1064nm (Experimental): Nd YAG laser 1064nm
  Interventions: Device: Nd YAG laser1064 nm
- combined two laser types (Experimental): combined fractional CO2 laser 10,600nm and Nd YAG laser 1064nm lasers treatment to keloid
  Interventions: Device: fractional CO2 laser 10,600nm; Device: Nd YAG laser1064 nm

INTERVENTIONS:
Device: fractional CO2 laser 10,600nm — fractional CO2 laser 10,600nm session, every month for 4 months
  Arms: combined two laser types; fractional CO2 laser 10,600nm
Device: Nd YAG laser1064 nm — Nd YAG laser1064 nm laser session, every month for 4 months
  Arms: Nd YAG laser 1064nm; combined two laser types

SUMMARY:
clinical comparative study comparing the effectiveness of fractional CO2, long pulsed Nd YAG and their combination in collagen remodeling in keloid clinically, biochemically and histopathologically

DETAILED DESCRIPTION:
Patients The study included 30 Egyptian patients with keloid scar recruited from the Out Patient Clinic, Dermatology Department, Cairo University.

Methodology

Patients:

- Thirty patients with keloid scar(s) were included in the study

- Every patient was subjected to the following:

1. Complete history taking: History of disease onset, course and duration, family history as well as history of any systemic or dermatological disease interfering with the eligibility of participation in the study.

   Thirty patients were included in the study which is a clinical comparative study comparing the effectiveness of fractional CO2, long pulsed Nd YAG and their combination in collagen remodeling in keloid clinically in all the included patients and biochemically and immunohistochemically fifteen patient
2. Full clinical examination:

   * General examination to determine any systemic or dermatological disease that might preclude the patient from participation in the study such as collagen disease.
   * Local examination to determine Fitzpatrick skin color of the patient and the site and extent of the scar to be treated.

   Methods:

   - Cases with multiple keloid scars three lesions 2 to 3 cm apart from each other were selected and labeled. The first one (lesion A) was treated using fractional CO2 laser 10,600 nm, the second (lesion B) long pulsed Nd YAG laser 1064 nm, while the last (lesion C) combined fractional CO2 followed by Nd YAG lasers after half an hour were used

   - patients who had a large sized lesion, the lesion was divided into three equal parts 2 to 3 cm apart from each other, they were labeled as areas A, B and C then subjected to the same treatment modalities as mentioned in case of multiple lesions.
   * Patients received 4 treatment sessions 4 to 8 weeks apart. Laser modalities and parameters
   * Topical anesthesia (lidocaine 2.5% and prilocaine 2.5%) was applied to the working area 30 to 60 minutes before the sessions, washed off and properly dried before the procedure.
   * Ablative fractional 10,600 nm carbon dioxide laser (DEKA smartxide DOT, Italy) and long pulsed Nd-YAG (DEKA synchro FT) were used in the treatment sessions with the following parameters Fractional CO2 Stacking: 5, Power: 20 Watt, Dwell time: 1000 micro second, Spacing : 800 micro meter fluence: 40 j/cm2 Pulse duration: 0.3 milli second Spot size: 5 mm Passes: 3.

   Assessment Assessment was done before treatment every session and one months after the final laser treatment. Clinical assessment was done for all patients while histopathological and biochemical assessment were done only in 15 patients.

   A. Clinical evaluation Clinical assessment was fulfilled via calculating the scores of both the Vancouver Scar Scale; and the Patient and Observer Scar Assessment Scale. Patients were assessed every session, any side effects were reported, e.g pain, swelling, infection, hyper pigmentation or hypo pigmentation.

   B. Histopathological and biochemical evaluation

   Fifteen patients were randomly selected and subjected to the pre and post treatment biopsies :
   * Pretreatment biopsy:

   Three mm punch skin biopsy was taken from the keloid (any lesion A, B, or C) before starting treatment sessions ●Post treatment biopsies: Each lesion (A, B, C) was biopsied separately (3 mm punch biopsy), one month after last treatment session.

   Biopsies of controls ●parts of excess skin from 12 patients undergoing abdominoplasty were used as controls for levels of TGFβ1 and TGFβ3.

   Procedure

   - Biopsies were fixed in 10 % neutral buffered formalin, and then embedded in paraffin blocks. Sections were prepared for routine staining by H&E. Other sections were prepared for histochemical staining of collagen fibres using Masson's trichrome stain and elastic fibres using orcein stain

   - All sections were examined using a Zeiss, Primo star light microscope (Zeiss, Germany). The microscope has an integrated camera by which photomicrographs depicting the various histopathological and histochemical findings were obtained. All photomicrographs presented in the thesis are according to their original magnification.

   • Evaluation of elastic fibres in orcein stained sections:

   Orcein stained sections were graded according to the grading criteria proved by Ozog et al. in 2013 for the appearance of the dermal elastic tissue as follows:

0 normal

1. short fragmented elastic fibres
2. intermediate between 1 and 3
3. fibrillar elastic fibres, parallel to epidermis
4. intermediate between 3 and 5
5. absent or nearly absent.

Image analyzer evaluation (morphometric study):

The area percent of collagen and elastic fibres were quantitatively evaluated in Masson's trichrome and orcein stained sections respectively at magnification X100 in 5 non overlapping fields for all patients. Image analysis was done using Leica Qwin 500C image analyzer computer system (England) present in the Histology Department, Faculty of Medicine, Cairo University .

ELIGIBILITY:
Inclusion Criteria:

* Patients with keloid scars of at least 6 months duration.
* No limitations regarding sex of the patients.
* Patients with three or more lesions 2 to 3 cm apart or patients having a large sized lesion.

Exclusion Criteria:

* Patients who had received any form of treatment during the last four weeks prior to treatment such as intralesional steroids or a laser procedure during the last six months.
* Patients with active skin infections e.g. herpes or autoimmune disease.
* Patients with previous history of adverse outcome related to laser therapy.
* Recent use of Isotretinoin (within 6 months prior to the procedure).
* Patients with known allergies to lidocaine.
* Smoking, pregnancy
* Patients with unrealistic expectations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
comparison between different laser modalities in treatment of keloids clinically | 5 months
  assessed by Patient and Observer Scar assessment Scale
comparison between different laser modalities in treatment of keloids morphometrically | 5 months
  assessed by Quantitative morphometric analysis using Leica Qwin 500 Image Analyzer (LEICA Imaging Systems Ltd, Cambridge, England) measuring area percent of collagen and elastin fibers in micrometer squared
comparison between different laser modalities in treatment of keloids biochemically | 5 months
  assessed by level of transforming growth factor beta 1 and 3 using Human TGF-B ELISA kit provided by ID labs Biotechnology London, ON, Canada.measurement unit is nano gram per gram tissue

CONTACTS AND LOCATIONS:
Overall Officials: Shereen O Tawfik, MD, Study Director — professor of Dermatology.faculty of medicine. Cairo university

IPD SHARING:
Plan to Share IPD: Undecided